CLINICAL TRIAL: NCT00814398
Title: Single Embryo Transfer Versus Double Embryo Transfer in Day 3 or Blastocyst Stage
Brief Title: Single Embryo Transfer Versus Double Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in cryopreservation protocol
Sponsor: Vida Recoletas Sevilla (Other)
Responsible Party: Principal Investigator, Manuel Fernandez-Sanchez, Primary Investigator, Vida Recoletas Sevilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IVISEV-002SET
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2011-03

CONDITIONS: Infertility
Keywords: Infertility; IVF; SET; DET; Blastocyst
MeSH Terms: conditions — Infertility | interventions — Single Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SET on day 3 (Experimental): Single embryo transfer on day 3 of embryo development
  Interventions: Procedure: Single Embryo Transfer (SET)
- DET on day 3 (Experimental): Double embryo transfer on day 3 of embryo development
  Interventions: Procedure: Double Embryo Transfer (DET)
- SET on day 5 (Experimental): Single embryo transfer on day 5 of embryo development
  Interventions: Procedure: Single Embryo Transfer (SET)
- DET on day 5 (Experimental): Double embryo transfer on day 5 of embryo development
  Interventions: Procedure: Double Embryo Transfer (DET)

INTERVENTIONS:
Procedure: Double Embryo Transfer (DET) — Two embryos are transferred during an IVF treatment
  Arms: DET on day 3; DET on day 5
Procedure: Single Embryo Transfer (SET) — A single embryo is transferred during an IVF treatment
  Arms: SET on day 3; SET on day 5

SUMMARY:
The aim of this project is to study the best number (1 or 2)and day (3 vs 5)of embryo transfer in good prognosis patient.

ELIGIBILITY:
Inclusion Criteria:G

* Good prognosis IVF patients

Exclusion Criteria:

* Bad prognosis IVF patients

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Live-birth delivery rate | End of pregnancy (nine months after last transfer)

SECONDARY OUTCOMES:
Multiple live-birth rate | End of pregnancy (nine months after last transfer)
Acceptance of assigned randomised group | Day of randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Fernandez, MD, Principal Investigator — Vida Recoletas Sevilla
Locations (1):
- IVI-Sevilla, Seville, Spain